CLINICAL TRIAL: NCT04982406
Title: Transcatheter Aortic Valve Replacement (TAVR) Effects on Cardiac Conduction System
Acronym: TAVR-HBE
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Alfred Buxton, Shlomo Ben-Haim, MD - Mark E. Josephson, MD, Professor of Medicine in Field of Cardiac Electrophysiology, Beth Israel Deaconess Medical Center
Other Study IDs: 2020P001189
Record Dates: First submitted 2021-07-20; First posted 2021-07-29 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Aortic Stenosis; Transcatheter Aortic Valve Replacement; Heart Block
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Block | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Transcatheter aortic valve replacement — Transcatheter aortic valve replacement

SUMMARY:
This is a prospective observational study, the purpose of which is to:

1. Characterize response of the AV conduction system to TAVR with various prostheses by recording continuous His bundle electrograms during valve placement.
2. Correlate preprocedure ECG features with changes in AV nodal and infranodal conduction during placement of the valve prosthesis.
3. Correlate changes in AV nodal and infranodal conduction during the procedure with risk of developing AV conduction block after TAVR.
4. Assess the contribution of stressing the conduction system by atrial pacing prior to and following TAVR to prediction of postprocedural heart block.

Assess the correlation between new onset bundle branch block, site and degree of conduction block or delay and subsequent development of high-grade or complete AV block.

DETAILED DESCRIPTION:
Study Population:

Inclusion criteria -all patients undergoing elective TAVR Exclusion criteria -patients with permanent implanted pacemakers or ICDs prior to TAVR

1. Record standard 12-lead ECG prior to procedure.
2. Place standard electrode catheter via a venous sheath prior to TAVR
3. Initially place the catheter in a proximal position with a large atrial electrogram and proximal His electrogram.
4. Record baseline His bundle electrogram. Record baseline AH and HV intervals.
5. Pace the atrium starting at a cycle length 100 ms shorter than the sinus cycle length, progressively reducing the paced cycle length in 20 ms decrements after 3 seconds pacing at each cycle length, while continuously monitoring arterial blood pressure, to A-V block.
6. Advance the distal electrodes while maintaining recording of a His bundle electrogram to a position where stable right ventricular pacing is secured. Record the RV pacing threshold.
7. If a stable right ventricular pacing position together with stable His bundle electrogram cannot be achieved, a second venous temporary pacing wire will be placed.
8. Record presence or absence of retrograde conduction during RV pacing at 4 times pacing threshold.
9. Ensure stable continuous His bundle electrogram recording while the aortic valve prosthesis is deployed.
10. Use the distal electrodes for rapid ventricular pacing at 4 times threshold during deployment of the valve prosthesis.
11. After the prosthesis has been deployed and is deemed stable, just prior to removing the RV catheter, record a final HBE (AH, HBE, SCL) and again pull back catheter to enable atrial capture with proximal electrodes - pace as above to AV block: start starting at a cycle length 100 ms shorter than the sinus cycle length, progressively reducing the paced cycle length in 20 ms decrements after 3 seconds pacing at each cycle length while monitoring continuous arterial blood pressure to A-V block.
12. Record 12-lead ECG after completion of the procedure and daily thereafter until hospital discharge.
13. Standard telemetry monitoring post procedure while hospitalized.
14. Upon hospital discharge place a standard continuous ambulatory ECG monitor for 2 weeks in patients that do not have a pacemaker implanted.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective TAVR at BIDMC

Exclusion Criteria:

* patients with permanent implanted pacemakers or ICDs prior to TA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe aortic stenosis or regurgitation planned to undergo transcatheter aortic valve replacement
Sampling Method: Non-Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Heart block | 30 days following procedure
  We will prospectively follow patients for the development of heart block requiring permanent pacemaker implantation, and identify factors associated with heart block following TAVR..

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Buxton, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Alfred Buxton, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Global Results will be published, not individual patient data

REFERENCES:
- [Result] Poulin MF, Ultimo B, Omar W, Rathakrishnan BG, Haouzi A, Pinto DS, Buxton AE, Laham RJ. Routine Electrophysiology Study During Transcatheter Aortic Valve Replacement: A Safety and Feasibility Pilot Study. JACC Cardiovasc Interv. 2023 Oct 23;16(20):2584-2586. doi: 10.1016/j.jcin.2023.07.017. Epub 2023 Sep 20. No abstract available. PMID 37737796